CLINICAL TRIAL: NCT06879522
Title: Feasibility and Early Efficacy of the Maximizing Energy Intervention for Decreasing Fatigue Impact in Breast Cancer Survivors
Brief Title: Maximizing Energy and Reducing Fatigue in Breast Cancer Survivors
Acronym: BCS_MAX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ketki Raina, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24050068
Record Dates: First submitted 2025-02-24; First posted 2025-03-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Survivor; Cancer Related Fatigue
Keywords: self-management; problem solving therapy; actigraphy; occupational therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximizing Energy (Experimental): Maximizing Energy
  Interventions: Behavioral: Maximizing Energy Intervention
- Health Education (Active Comparator): Health Education
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Maximizing Energy Intervention — A licensed occupational therapist will deliver the intervention. The Maximizing Energy program combines problem-solving therapy (PST) and energy conservation education. Participants will participate in 6 virtual once/week sessions for 30 minutes. The introductory session, they will track their fatigue and identify three key fatigue-related problems. In session 2, they will prioritize one problem and practice problem-solving steps. They then implement an action plan and review progress in the next session. If the solution is ineffective, the therapist helps modify it or create a new one. If successful, the participant moves to the next problem. A MAX workbook supports learning, covering intervention details, fatigue education, energy conservation strategies, and problem-solving worksheets. The goal is to help participants apply these strategies to improve daily life and return to work.
  Arms: Maximizing Energy
Behavioral: Health Education — To control for the effects of interactions with an interventionist, participants in the attention control group will receive the Health Education intervention. The interventionists will review a workbook covering fatigue, energy conservation, healthy eating, exercise, and relaxation. Like the MAX intervention, Health Education will be delivered virtually in weekly 30-minute one-on-one sessions for six weeks. The interventionist provides education on breast cancer-related fatigue, diet, safe physical activities, and energy conservation strategies tailored to individual needs. A workbook will support learning.
  Arms: Health Education

SUMMARY:
This study is testing a program called Maximizing Energy to see if it can help women who have finished breast cancer treatment manage their fatigue. The study has two main goals:

1. Check if the program can be successfully delivered - Researchers will see if women are willing to join and stay in the study, if they follow the program, and if they find it helpful.
2. See if the program works - Researchers will compare Maximizing Energy to a general health education program to see which one helps reduce cancer-related fatigue better.

Participant will:

1. Take tests to see if they qualify and to measure their fatigue.
2. Be randomized to receive Maximizing Energy or Health Education Interventions for 6 sessions over the internet
3. After the sessions and again one month later, repeat some tests to see if their fatigue has improved.

ELIGIBILITY:
Inclusion Criteria:

* adult (18 years and older) pre and post-menopausal female at birth diagnosed with Stages I-IIIa breast cancer,
* completed primary treatment for breast cancer (surgery, chemotherapy, radiation) at least 6 months prior to ensure that fatigue is stable and chronic, - moderate to severe fatigue based on score ≥ 4 on the 7-point Fatigue Severity Scale,
* able to speak and understand English
* has a mobile device that runs on the Apple or Android platform

Exclusion Criteria:

* major depressive disorder, mania, hypomania, psychosis, or substance abuse in the past 3 months and
* disability due to diagnoses other than breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Retention in the study | Baseline to Week 11 (4 weeks post-intervention)
  The proportion of participants who remain in the study until its completion relative to those initially enrolled.
  The retention rate will be calculated separately for the Maximizing Energy and Control Groups using the following formula: (number of participants who completed the study/number of participants initially enrolled)X 100
Participant Adherence to treatment: Receipt | Week 7 (post-6-week intervention)
  The investigators will collect data on the number of intervention sessions attended by participants
Participant Adherence to treatment: Receipt | Week 7 (post-6-week intervention)
  Interventionists will rate participant's active engagement in the interventions on the Pittsburgh Participant Rating Scale. Each session will be scored 1 (no engagement, refusal) to 6 (excellent engagement) by the interventionist conducting the sessions.
Participant Adherence to treatment: Enactment | Week 7(post-6-week intervention)
  The investigators will collect interventionist rating of whether participant completed action plan from previous session (3-point scale; 0 = not completed, 2 = plan completed) for the MAX Intervention group only.
Participant Satisfaction with Intervention | Week 7(post-6-week intervention)
  Client satisfaction is measured using the Client Satisfaction Questionnaire. The Clients Satisfaction Questionnaire is an 8-item assessment of satisfaction with the intervention program, rated on a 4-point scale that ranges from 1 to 4 in each item. Higher scores indicate greater satisfaction with the intervention.
Intervention Fidelity | Week 7(post-6-week intervention)
  All intervention sessions will be video recorded and a random 20 percent will be rated by independent evaluators trained by the principal investigator. Intervention fidelity for both groups will be assessed using the PST Provider Checklist. The a priori criterion for adequate fidelity was that equal or greater than 80 percent of intervention sessions are rated with equal or greater than 80 percent of adequate fidelity for the MAX Intervention group while less than 20 percent of intervention sessions are rated with equal or lesser than 20 percent of adequate fidelity for the Health Education group.
Changes in fatigue | Baseline to Week 11 (4 weeks post-intervention)
  The PROMIS® Item Bank v1.0 - Fatigue - Short Form 13a (FACIT-Fatigue) is a 13-item questionnaire designed to assess fatigue levels and their impact on daily activities and quality of life. Each item is scored on a 5-point Likert scale (1 = not at all to 5 = very much), with a total score ranging from 13 to 65. Higher scores indicate greater fatigue, while lower scores suggest less fatigue and better energy levels.

SECONDARY OUTCOMES:
Changes in resilience | Baseline to Week 11 (4 weeks post-intervention)
  The Connor-Davidson Resilience Scale (CD-RISC) is a tool designed to measure an individual's resilience, or ability to adapt to stress and adversity. It consists of 25 items, each rated on a 5-point Likert scale (0 = not true at all to 4 = true nearly all the time), with total scores ranging from 0 to 100. Higher scores indicate greater resilience, reflecting stronger coping skills and adaptability in challenging situations.
Changes in impact of fatigue in daily life | Baseline to Week 11 (4 weeks post-intervention)
  The Modified Fatigue Impact Scale (MFIS) is a 21-item questionnaire that assesses the impact of fatigue on physical, cognitive, and psychosocial functioning. Each item is rated on a 5-point Likert scale (0 = never to 4 = almost always), with a total score ranging from 0 to 84. Higher scores indicate a greater negative impact of fatigue on daily life, while lower scores suggest minimal interference with functioning.
Changes in fatigue severity | Baseline to Week 11 (4 weeks post-intervention)
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire designed to assess the impact of fatigue on daily life and functioning. Each item is rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with total scores ranging from 9 to 63. Higher scores indicate greater fatigue severity and its interference with daily activities, while lower scores suggest minimal fatigue impact.
Change in physical activity: Step Count | Baseline to Week 11 (4 weeks post-intervention)
  The investigators will collect data on physical activity as a surrogate measure of increase in energy. The ActiGraph wGT3X-BT® is a validated accelerometer used to measure physical activity outcomes, including step count. The ActiGraph wGT3X-BT will be worn on the wrist for 5 days to yield three 24 hour data for a mean number of steps taken daily.
Change in Physical Activity: Energy Expenditure | Baseline to Week 11 (4 weeks post-intervention)
  The investigators will collect data on physical activity as a surrogate measure of increase in energy. The ActiGraph wGT3X-BT® is a validated accelerometer used to measure physical activity outcomes, including energy expenditure. The ActiGraph wGT3X-BT will be worn on the wrist for 5 days to yield three 24 hour data for a mean energy expenditure daily.
Change in physical activity: Intensity of Activity | Baseline to Week 11 (4 weeks post-intervention)
  The investigators will collect data on physical activity as a surrogate measure of increase in energy. The ActiGraph wGT3X-BT® is a validated accelerometer used to measure physical activity outcomes, including percentage of time spent in sedentary, light, moderate, and vigorous physical activity. The ActiGraph wGT3X-BT will be worn on the wrist for 5 days to yield three 24 hour data for a percentage of time spent in different intensity activity daily.

OTHER OUTCOMES:
Commonly used strategies to manage fatigue | Baseline to 4-weeks after intervention completion
  The Energy Conservation Strategies Survey assesses which energy conservation strategies they have used in the past 6 weeks and how effective they perceive these strategies to be in managing their fatigue. The survey lists 14 strategies. Strategy effectiveness in managing fatigue is rated on a 10-point scale with 1 indicating not effective and 10 indicating very effective.

CONTACTS AND LOCATIONS:
Overall Officials: Ketki Raina, PhD, OTR/L, FAOTA, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No